CLINICAL TRIAL: NCT01818778
Title: The Efficacy of Using Volunteers to Implement a Cognitive Stimulation Program in Two Long-Term Care Homes
Acronym: VolCogStim
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Baycrest (Other)
Responsible Party: Principal Investigator, Dr. John Kirby, Ph.D., Queen's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Queens-Baycrest 65
Record Dates: First submitted 2013-03-19; First posted 2013-03-26 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Impaired Cognition; Geriatric Disorder; Learning Disorders; Age-Related Memory Disorders; Impairment of Attention
MeSH Terms: conditions — Cognition Disorders; Learning Disabilities; Memory Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stimulation Group (Experimental): Cognitive Stimulation Group: One-on-one (one volunteer visiting one resident at a time), stimulation-group residents and stimulation-group volunteers met 3 times each week, for 8 weeks, to work through a variety of memory, reasoning, and selective attention exercises. Each visit was 20 minutes in length.
  Interventions: Other: Cognitive stimulation program
- Control Group (Active Comparator): Standard "Friendly Visit": Control-group residents and control-group volunteers, one-on-one, met for 8 weeks, 3 times each week, for "friendly visits". Each visit was 20 minutes in length.
  Interventions: Other: Standard Friendly Visit

INTERVENTIONS:
Other: Cognitive stimulation program — The stimulation program was composed of therapy- and education-based exercises which were specifically designed to stimulate reasoning, memory, and attention skills in adults.
  Arms: Stimulation Group
Other: Standard Friendly Visit — Volunteers provided standard "friendly visits" to residents which included a friendly greeting and casual conversation about issues which interest the resident.
  Arms: Control Group

SUMMARY:
Many volunteers visiting seniors make socially-based "friendly visits". This study investigated the efficacy of volunteers making visits focused on stimulating cognition. Participants were randomly assigned to either a "friendly visit" control group or a cognitive stimulation group. Seniors receiving stimulation visits made statistically significant improvement in memory abilities.

DETAILED DESCRIPTION:
Older adults who maintain their cognitive skills and abilities are able to live more independently than those whose skills have deteriorated. The costs (money, time, personnel) associated with providing cognitive stimulation programs to residents in long-term care homes often prohibit the delivery of these programs. The present study explored the efficacy of using volunteers to administer a stimulation program in two long-term care homes. The program focused on stimulating reasoning, attention, and memory abilities using uncomplicated, pen-and-paper exercises. Thirty-six resident participants and 16 volunteer participants were randomly assigned to one of two parallel groups, either the control or stimulation group.

For eight weeks, three times each week, control group participants met for standard "friendly visits" (casual conversation between a resident and volunteer) and stimulation group participants met to work through a variety of exercises meant to stimulate the cognitive abilities of residents. Results were analyzed using a 2-way ANOVA and indicated statistically significant Group x Time interactions for Verbal Memory (F(1, 33) = 7.92, p = .008), Non-Verbal Memory (F(1, 33) = 6.8, p = .014), Learning (F(1, 33) = 5.27, p = .028), and Verbal Fluency (F (1, 33) = 5.56, p = .024).

Volunteers completed a post-study questionnaire which indicated that the volunteers in the stimulation group found their skills-based interactions more stimulating for residents. Given this showing of improved resident abilities, it is reasonable to assert that the study does demonstrate that a volunteer-administered, cognitive stimulation program can provide measurable gains in the cognitive abilities of older adults. Further studies concerning the role of volunteers in the maintenance of the cognitive abilities of older adults are recommended.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and over
* living in a long-term care home
* normal or corrected visual and auditory acuity
* English proficiency
* not currently using de-stabilizing, psychotropic medication known to impair cognition
* ability and willingness to actively listen to and accurately follow 2-step instructions for at least 20 consecutive minutes

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Test of Memory and Learning - Senior Edition (TOMAL-SE) | 10 weeks
  The TOMAL-SE was designed specifically for seniors and provides a thorough assessment, without being fatiguing (Reynolds & Vorees, 2012). The battery includes normative data for ages 55:0-89:11. It is a paper-based test and takes approximately 25-35 minutes to administer. It provides scores for the following indexes: Verbal Memory, Non-Verbal Memory, Delayed Memory, and Learning.

SECONDARY OUTCOMES:
Wechsler Abbreviated Scale of Intelligence - Second Edition (WASI-II; Wechsler, 2011) | 10 weeks
  The WASI-II is designed to measure intelligence. The latest version, published in 2011, includes normative data for ages 6:0-90:11 years. The paper-based, two-subtest form includes the Vocabulary and Matrix Reasoning tests and provides an estimate of general cognitive ability.

OTHER OUTCOMES:
Letter Sorting Test | 10 weeks
  This test assesses working memory and concentration. Participants were asked to spell a 5-digit word, forwards, backwards, and in alphabetical order. To score the test, 1 point each was given for spelling the word correctly forwards, backwards and in alphabetical order. The test usually took approximately 2 minutes to administer.
Clock Drawing Test | 10 weeks
  In this test, participants were given a sheet of paper with a circle on it. They were then be asked to follow a two-step instruction: "This is a clock. Please draw all the numbers on it and the time 'ten past eleven'". This test was originally developed to assess visuo-constructional abilities, but it also requires language comprehension, numerical knowledge, strategy planning, and memory. To score the test, the 6-point Shulman et al. (1993) scoring method will be employed where higher scores reflect a greater number of errors and more impairment. The test took approximately 2 minutes to complete.
Action "Verbal Fluency" Test | 10 weeks
  A test of action verbal fluency was applied to measure working memory, planning, organization, and word retrieval. Residents were asked to generate as many action words, in their infinitive form (i.e., eat, smell, etc.) as possible within 60 seconds. One point was given for each action word stated. Verbal instructions explicitly stated that no points would be awarded for the use of the same word with different endings, like eat, eating, and eaten. The test took approximately 1-2 minutes to administer.

CONTACTS AND LOCATIONS:
Overall Officials: John Kirby, Ph.D., Principal Investigator — Queen's University
Locations (1):
- Baycrest, Toronto, Ontario, Canada